CLINICAL TRIAL: NCT00408356
Title: Immunological and Clinical Responses to Zinc: A Randomized, Double-Blind Trial of Zinc Treatment vs. Zinc Treatment Plus Daily Supplementation for 3 Months Among Children Under 2 Years of Age With an Acute Diarrheal Illness.
Brief Title: Immunological and Clinical Responses to Zinc in Children With Diarrhoea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Dr. Firdausi Qadri, International Centre for Diarrhoeal Diseases Research, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2004-017
Record Dates: First submitted 2006-12-05; First posted 2006-12-06 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Diarrhoea
Keywords: Zinc treatment; supplementation; Enterotoxigenic E. coli; diarrhoea
MeSH Terms: conditions — Diarrhea | interventions — Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Zinc

SUMMARY:
Zinc deficiency has been found to be widespread among children in developing countries.Clinical and field studies have consistently observed an association between zinc deficiency and higher rates of infectious diseases, including skin infections, diarrhea, respiratory infections, malaria, and delayed wound healing. Based upon the impact of zinc deficiency on diarrheal disease alone, it is estimated correction of this deficiency could save 450,000 under-five deaths annually. What is the physiological explanation for this? Zinc has been identified to play critical roles in metallo-enzymes, poly-ribosomes, the cell membrane, and cellular function, leading to the understanding that it also plays a central role in cellular growth and in the function of the immune system. With zinc deficiency epithelial barriers are compromised and multiple components of the immune system malfunction. The obvious conclusion is that zinc deficiency results in diminished immunological competence that in turn leads to an increased risk for infectious diseases and greater severity of illnesses. Whether this is the case requires substantiation. A related, but more pragmatic question is the value added of zinc supplementation in addition to zinc treatment. The scale-up strategy being pursued in Bangladesh is to provide zinc for 10 days as a treatment at the time of a diarrhea episode. This is in accordance with recently revised WHO recommendations for the treatment of childhood diarrhea (WHO, in press). Can we conclude there is no or minimal value added to continuing zinc as a dietary supplement in zinc deficient children following an acute episode? If there is added benefit, can this be explained by improvement in zinc levels and/or immune function? The aims of this study include:1. In children six to twenty-four months of age with an acute episode of diarrhea attributable to enterotoxigenic E. coli (ETEC), to describe the innate and adaptive immune response to zinc and to relate changes in immune function or zinc status to the occurrence of repeat infectious illnesses over a 9 month period of observation. 2a. In children six to twenty-four months of age with an acute episode of diarrhea with enterotoxigenic E. coli (ETEC), and other non-ETEC diarrhea, to determine the value added of zinc supplementation following treatment in terms of the future occurrence of ACD, ARI, and impetigo and 2b. to assess the impact of zinc supplementation on health services utilization and household expenditures for ACD, ARI and impetigo.

ELIGIBILITY:
Inclusion Criteria:

* Children 6-24 months of age with acute childhood diarrheal illness.

Exclusion Criteria:

* Severe dehydration, suspected cholera or pneumonia, chronic illness, bipedal edema (seriously ill children will be referred to ICDDR,B/Shishu Hospital).
* The child is currently receiving zinc (as a treatment or supplement)
* Wt/length, z-score below -3 (these children will be referred to ICDDR,B/ Shishu Hospital)
* Already participating in another study involving nutritional or therapeutic interventions

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 338 (Estimated)
Dates: Start 2004-11; Primary Completion 2006-08 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To evaluate innate and adaptive immune response.
Future occurrence of acute diarrhoea, ARI and impetigo.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Saha, MBBS, Study Director — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- ICDDR,B. Mirpur Field Site, Dhaka, Bangladesh

REFERENCES:
- [Derived] Sheikh A, Shamsuzzaman S, Ahmad SM, Nasrin D, Nahar S, Alam MM, Al Tarique A, Begum YA, Qadri SS, Chowdhury MI, Saha A, Larson CP, Qadri F. Zinc influences innate immune responses in children with enterotoxigenic Escherichia coli-induced diarrhea. J Nutr. 2010 May;140(5):1049-56. doi: 10.3945/jn.109.111492. Epub 2010 Mar 17. PMID 20237063